CLINICAL TRIAL: NCT07300215
Title: An Exploratory Study on Individualized Neoadjuvant Treatment Regimens for Early HR+/HER2+ Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Bengbu Medical University (Other)
Responsible Party: Principal Investigator, Gongsheng, Jin, chief physicians, The First Affiliated Hospital of Bengbu Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025KY060
Record Dates: First submitted 2025-12-10; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental)
  Interventions: Drug: individualized neoadjuvant treatment

INTERVENTIONS:
Drug: individualized neoadjuvant treatment — For HR+/HER2+ breast cancer patients treated with TCbHP, after 2 cycles of treatment, they were classified according to the therapeutic effect into the effective group and the group without early response. The effective group continued to receive TCbHP treatment for another 4 cycles, while the group without early response changed to the neoadjuvant treatment regimen of trastuzumab dual-target combined with exemestane and palbociclib for 4 cycles.
  Evaluation methods:
  Early non-response is defined as the results of the examination after the end of the 2nd cycle of treatment meeting any of the following criteria:
  1. MRI, ultrasound: PD/SD of lymph nodes or primary lesion, PR but tumor regression < 50%;
  2. Histological pathological examination:Changes in immunohistochemical molecular typing;The decrease in Ki-67 compared to the baseline is less than 20%;PIK3CA mutation.

SUMMARY:
HR+/HER2+ breast cancer belongs to a special type of tumor with dual-channel signal activation. However, in clinical treatment, the preferred approach is usually the inhibition of the HER2 signaling pathway. Therefore, the non-pCR rate after neoadjuvant therapy is relatively high (about 60%). To optimize the neoadjuvant treatment strategy for HR+/HER2+ breast cancer, increase the pCR rate of neoadjuvant treatment, and improve the prognosis of patients, our research group intends to conduct a prospective clinical and translational study. By observing the clinical efficacy and changes in biomarkers, individualized treatment for HR+/HER2+ breast cancer will be carried out. Patients who respond well to HER2-targeted therapy will be identified early, and for those without early relief, targeted combined dual-channel inhibition therapy with endocrine treatment will be adopted. The effectiveness and safety of the individualized neoadjuvant treatment strategy for HR+/HER2+ breast cancer patients will be evaluated. In addition, this study aims to focus on the neoadjuvant chemotherapy mechanism of HR+/HER2+ breast cancer, and combine the establishment and validation of effective disease models to provide theoretical basis and experimental support for achieving precise treatment and clinical transformation.

ELIGIBILITY:
Inclusion Criteria:

* The patient must meet all of the following criteria to be included in the study:

  1. The tumor stage must be in accordance with the 8th edition of the AJCC standard, being stage II-III for the initial diagnosis;
  2. The age must be between 18 and 75 years (inclusive of 18 and 75), and the patient must be female;
  3. All patients must have been pathologically confirmed as HR+/HER2+. The estrogen receptor (ER) must be positive (>10%) or the progesterone receptor (PR) must be positive (>10%), and the HER2 must be positive. HER2 positivity is defined as an immunohistochemistry (IHC) score of 3+, or a score of 2+ and positive in in situ hybridization (ISH) (ISH amplification rate ≥ 2.0);
  4. The ECOG score must be 0-1;
  5. According to the RECIST 1.1 standard, there must be at least one measurable lesion;
  6. The functional levels of the organs must meet the following requirements: (a) Blood routine: ANC ≥ 1.5×109/L; PLT ≥ 90×109/L; Hb ≥ 90g/L; (b) Blood biochemistry: TBIL ≤ 1.5×ULN; ALT and AST ≤ 3×ULN; BUN and Cr ≤ 1.5×ULN and creatinine clearance rate ≥ 50 mL/min; (c) Cardiac echocardiography: Left ventricular ejection fraction ≥ 50%:
  7. The subject voluntarily joins this study, signs the informed consent, has good compliance and is willing to cooperate with follow-up.

Exclusion Criteria:

* (1) Has received any form of anti-tumor treatment (chemotherapy, radiotherapy, molecular targeted therapy, endocrine therapy, etc.) in the past; (2) Is currently receiving other anti-tumor drug treatment; (3) Has had any other malignant tumor within the past 5 years, except for cured cervical carcinoma in situ, basal cell carcinoma or squamous cell carcinoma of the skin, or minimally invasive papillary thyroid cancer after radical surgery; (4) Has severe dysfunction of important organs such as the heart, liver, and kidneys; (5) Has difficulty swallowing, chronic diarrhea, and intestinal obstruction, and has multiple factors that affect the administration and absorption of the drugs; (6) Has participated in other drug clinical trials within 4 weeks before enrollment and has received the investigational drugs; (7) Has a history of immunodeficiency diseases, including positive HIV test, HCV, active viral hepatitis, or having other acquired or congenital immune deficiency diseases, or having a history of organ transplantation; (8) Has a known history of allergic reaction to the components of this study drug; (9) Has had any heart disease, including: requiring drug treatment or clinically significant arrhythmia; myocardial infarction; heart failure; any other heart disease judged by the investigator as unsuitable for participation in this trial; (10) Pregnant or lactating female patients, female patients with reproductive capacity and positive baseline pregnancy test results; (11) According to the investigator's judgment, has serious accompanying diseases that endanger the patient's safety or affect the patient's completion of the study (including but not limited to severe hypertension that cannot be controlled by drugs, severe diabetes, active infection, etc.); (12) Has a clear history of neurological or mental disorders, including epilepsy or dementia; (13) The investigator deems that the patient is not suitable for participating in this study in any other circumstances.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
tpCR rate，total physiological complex response | From the time of enrollment to one month after the surgery
  After the resection of the primary tumor, microscopic examination of the breast and the ipsilateral axillary lymph nodes revealed no invasive tumor cells (ypT0/is ypN0)

SECONDARY OUTCOMES:
bpCR，breast physiological complex response | From the time of enrollment to one month after the surgery
  After the primary tumor was removed, microscopic examination of the breast revealed no invasive tumor cells (ypT0/is)
EFS，Event-free survival | baseline，1year，up to 2year
  The time from the start of medication to the occurrence of any of the following events for the first time: disease progression making surgical treatment impossible, local or distant recurrence, death due to any cause, etc.
ORR，Objective Response Rate | 6-12 months
  The proportion of patients whose tumor volume has decreased by 30% and has remained stable for more than four weeks is referred to as the sum of complete response (CR) and partial response (PR).
OS，Overall Survival | baseline，1year，up to 2year
  Refers to the period from the start of medication use until death occurs due to any cause.
adverse event | up to 2year
  Collect all adverse events that occurred in all subjects from the signing of the informed consent to 28 days after the cessation of medication, including clinical symptoms and abnormal vital signs, as well as abnormalities in laboratory tests. Record the clinical manifestations, severity, occurrence time, duration, treatment methods, prognosis, and determine the correlation between these events and the test drug.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol